CLINICAL TRIAL: NCT05410821
Title: An Open-Label, Non-Randomized, Dose Escalation, Single-Center, Investigator-Initiated Trial to Determine the Safety, Dosimetry, and Preliminary Effectiveness of 177Lu-DOTA-EB-FAPI in Metastatic Radioactive Iodine Refractory Thyroid Cancer Patients With Progressive Disease After Tyrosine Kinase Inhibitors Treatment
Brief Title: Evaluation of 177Lu-DOTA-EB-FAPI in Patients With Metastatic Radioactive Iodine Refractory Thyroid Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XMYY-2022KY054
Record Dates: First submitted 2022-06-05; First posted 2022-06-08 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Refractory Thyroid Gland Carcinoma; Refractory Thyroid Gland Papillary Carcinoma; Refractory Thyroid Gland Follicular Carcinoma; Refractory Thyroid Gland Hurthle Cell Carcinoma
Keywords: radioactive iodine refractory thyroid cancer; RAIR-TC; radioligand therapy; 177Lu-DOTA-EB-FAPI
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Cancer, Papillary; Adenocarcinoma, Follicular; Thyroid cancer, Hurthle cell

STUDY DESIGN:
Intervention Model Description: classic 3+3 dose escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 177Lu-DOTA-EB-FAPI 1 (Experimental): 177Lu-DOTA-EB-FAPI A maximum of 2 cycles of 60 mCi (2.22 GBq) 177Lu-DOTA-EB-FAPI, each. Route of administration: Slow intravenous infusion/injection (i.v.) Duration of treatment: 2 cycles, every 6 weeks
  Interventions: Drug: 177Lu-DOTA-EB-FAPI 1 radionuclide therapy
- 177Lu-DOTA-EB-FAPI 2 (Experimental): 177Lu-DOTA-EB-FAPI A maximum of 2 cycles of 90mCi (3.33 GBq) 177Lu-DOTA-EB-FAPI, each. Route of administration: Slow intravenous infusion/injection (i.v.) Duration of treatment: 2 cycles, every 6 weeks
  Interventions: Drug: 177Lu-DOTA-EB-FAPI 2 radionuclide therapy
- 177Lu-DOTA-EB-FAPI 3 (Experimental): 177Lu-DOTA-EB-FAPI A maximum of 2 cycles of 135 mCi (4.99 GBq) 177Lu-DOTA-EB-FAPI, each. Route of administration: Slow intravenous infusion/injection (i.v.) Duration of treatment: 2 cycles, every 6 weeks
  Interventions: Drug: 177Lu-DOTA-EB-FAPI 3 radionuclide therapy

INTERVENTIONS:
Drug: 177Lu-DOTA-EB-FAPI 1 radionuclide therapy — radionuclide therapy using 177Lu-DOTA-EB-FAPI 60 mCi (2.22 GBq) will be performed 6-weekly. A maximum of 2 cycles will be administered.
  Arms: 177Lu-DOTA-EB-FAPI 1
Drug: 177Lu-DOTA-EB-FAPI 2 radionuclide therapy — radionuclide therapy using 177Lu-DOTA-EB-FAPI 90 mCi (3.33 GBq) will be performed 6-weekly. A maximum of 2 cycles will be administered.
  Arms: 177Lu-DOTA-EB-FAPI 2
Drug: 177Lu-DOTA-EB-FAPI 3 radionuclide therapy — radionuclide therapy using 177Lu-DOTA-EB-FAPI 135 mCi (4.99 GBq) will be performed 6-weekly. A maximum of 2 cycles will be administered.
  Arms: 177Lu-DOTA-EB-FAPI 3

SUMMARY:
Increased fibroblast activation protein expression is positively correlated with the dedifferentiation and aggressiveness of thyroid cancer. Radiolabeled fibroblast activation protein inhibitor therapy, also known as radioligand therapy has become a novel treatment for patients with radioactive iodine refractory thyroid cancer and disease progression after first-line treatment. However, a major problem in the therapeutic use of 177Lu-DOTA-FAPI has been its short half-life and fast rate of clearance. This study was designed to evaluate the safety, tolerability, and maximum tolerated dose of a long-lasting radiolabeled fibroblast activation protein inhibitor 177Lu-DOTA-EB-FAPI in mRAIR-TC patients with PD after TKIs treatment.

DETAILED DESCRIPTION:
This dose-escalation study will include a maximum of 20 mRAIR-TC subjects with progressive disease after tyrosine kinases inhibitors (TKIs) treatment, with an increased radiotracer uptake in tumors on 68Ga-FAPI-46 PET/CT. The initial dose of 177Lu-DOTA-EB-FAPI is 2.22GBq (60 mCi), and subsequent cohorts receive an incremental 50% dose increase until dose-limiting toxicity (DLT) was observed. Treatment is planned for up to 2 cycles, and the time interval between cycles is 6 weeks. The primary endpoint assessed the safety and maximum tolerated dose of 177Lu-DOTA-EB-FAPI used for radioligand therapy in patients with advanced mRAIR-TC. Secondary endpoints included dosimetry and determination of the preliminary treatment efficacy of 177Lu-DOTA-EB-FAPI.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign a written informed consent document.
2. Age 18 and older
3. Confirmed unresectable or metastatic radioactive iodine refractory thyroid cancer with measurable disease per RECIST (version 1.1) (i.e. at least 1 lesion > 1 cm or lymph node > 1.5 cm in short axis)
4. Progressive disease after TKIs treatment
5. Eastern Cooperative Oncology Group Performance Status ≤ 3
6. Participant must have completed prior therapy at least 2 weeks (washout period) prior to 68Ga-FAPI-46 PET/CT scan. Any clinically significant toxicity (with the exceptions of hair loss and sensory neuropathy) related to prior therapy resolved below Grade 2 or baseline. Completion of entry into 68Ga-FAPI-46 study and completion of scan
7. Hematologic parameters defined as:

Absolute neutrophil count (ANC) ≥ 1000 cells/mm3 Platelet count ≥ 50,000/mm3 Hemoglobin ≥ 8 g/dL

Blood chemistry levels defined as:

AST, ALT, alkaline phosphatase ≤ 5 times upper limit of normal (ULN) Total bilirubin ≤ 3 times ULN Creatinine ≤ 3 times ULN Able to remain motionless for up to 30-60 minutes per scan

Exclusion Criteria:

1. Participant on any chemical anticoagulant including antiplatelet agents (excluding ASA)
2. Participants with Class 3 or 4 NYHA Congestive Heart Failure
3. Clinically significant bleeding within two weeks prior to trial entry (e.g. gastrointestinal bleeding, intracranial bleeding)
4. Pregnant or lactating women
5. Major surgery, defined as any surgical procedure that involves general anesthesia and a significant incision (i.e. larger than what is required for placement of a central venous access, percutaneous feeding tube, or biopsy) within 28 days prior to study day 1 or anticipated surgery within the subsequent 6 weeks
6. Has an additional active malignancy requiring therapy within the past 2 years
7. Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy
8. Psychiatric illness/social situations that would interfere with compliance with study requirements
9. Cannot undergo PET/CT scanning because of weight limits (350 lbs)
10. INR>1.2; PTT>5 seconds above UNL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events (safety and tolerability) | From date of involvement until 6 weeks after the second treatment cycles
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0. Dose-limiting toxicity was defined as any 177Lu-DOTA-EB-FAPI-related AE ≥ grade 3 (G3).
To determine the maximum tolerated dose (MTD) | From date of involvement until 6 weeks after the second treatment cycles
  The MTD is the dose level below that which 2 out of 6 subjects in a cohort have DLT

SECONDARY OUTCOMES:
Objective response rate (ORR) | baseline, 6 weeks after each treatment cycle
  68Ga-Fibroblast activation protein inhibitor 46 will be performed for efficacy evaluation by RECIST 1.1. Particularly, 68Ga-FAPI-46 will be performed at baseline, and 6 weeks after each treatment cycle.
Dosimetry | Dosimetry was estimated in the first treatment cycle for each patient
  Dosimetry, measured as absorbed dose in tumor and normal organs (Gy/GBq), was estimated in the first treatment cycle for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Haojun Chen, MD, PhD, Study Chair — The First Affiliated Hospital of Xiamen University
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, China

IPD SHARING:
Plan to Share IPD: No